CLINICAL TRIAL: NCT06600243
Title: Could Microfiltered-seawater Supplementation and Variable Resistance Training Improve Blood Pressure, Oxidative Stress, Hepatic, and Renal Biomarkers in Older Women? a 32-week, Double-blinded, Randomized, Placebo-controlled Trial
Brief Title: Influence of Microfiltered-seawater Supplementation and Variable Resistance Training in Blood Pressure, Oxidative Stress, Hepatic, and Renal Biomarkers in Older Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Juan C. Colado, Professor, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: H1414072784009
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Blood Pressure; Oxidative Stress; Renal Disease; Hepatic Impairment
Keywords: aged; postmenopause; bone mineral density; muscle strength
MeSH Terms: conditions — Kidney Diseases | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Resistance training + deep sea water (Experimental): Resistance training with elastic bands prior intake of deep sea water (20ml) twice weekly during 32 weeks.
  Interventions: Dietary Supplement: Resistance training + deep sea water
- Resistance training + Placebo (Active Comparator): Resistance training with elastic bands prior placebo water (20ml) twice weekly during 32 weeks.
  Interventions: Dietary Supplement: Resistance training + Placebo
- Control + Deep sea water (Active Comparator): No exercise and intake of deep sea water (20ml) twice weekly during 32 weeks.
  Interventions: Dietary Supplement: Control + deep sea water
- Control + Placebo (Placebo Comparator): No exercise and intake of placebo water (20ml) twice weekly during 32 weeks.
  Interventions: Dietary Supplement: Control + Placebo

INTERVENTIONS:
Dietary Supplement: Resistance training + deep sea water — A group that will perform a resistance training protocol with variable resistance and at the same time will receive a supplementation composed by deep sea water
  Arms: Resistance training + deep sea water
Dietary Supplement: Resistance training + Placebo — A group that will perform a resistance training protocol with variable resistance and at the same time will receive a placebo supplementation that have the same tasted than the deep sea water supplementation
  Arms: Resistance training + Placebo
Dietary Supplement: Control + deep sea water — A group that will maintain their usual live and at the same time will receive a supplementation composed by deep sea water
  Arms: Control + Deep sea water
Dietary Supplement: Control + Placebo — A group that will maintain their usual live and at the same time will receive a placebo supplementation that have the same tasted than the deep sea water supplementation
  Arms: Control + Placebo

SUMMARY:
This study was conducted to investigate the effects of the intake of deep sea water prior to resistance training on blood pressure, oxidative stress and hepatic and renal variables in older women.

DETAILED DESCRIPTION:
This study was a 32 weeks, double-blinded, randomized, placebo-controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* (i) women aged ≥65years
* (ii) able to climb 10 stairs without pause and walk 100m without a walker
* (iii) score above 23 points in the mini-mental state examination
* (iv) <1h of physical activity per week throughout the six months before the study
* (v) possess a medical certificate of aptitude to carry out physical activity

Exclusion Criteria:

Participants who had suffered:

* (i) any type of musculoskeletal, cardiovascular, hepatic, renal, pulmonary, neurological, or neuromuscular injury or disorder and/or
* (ii) taking any type of drug/supplement that may alter the results of the study (e.g., vitamin C, vitamin E, estrogens, beta-blockers, calcitonin, steroid hormones, etc.)
* (iii) changes in body weight of more than 10% in the year prior to the study
* (iv) have a severe hearing or visual impairment
* (v) participate in another research project (within the last six months) involving an exercise, dietetic and/or pharmaceutical intervention

Min Age: 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 109 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Malondialdehyde (MDA) | pre (week 0) and post (week 32)
  Oxidative stress biomarker
Oxidized/reduced glutathione ratio (GSH/GSSG) | pre (week 0) and post (week 32)
  Antioxidant enzyme
Interleukin-6 (IL-6) | pre (week 0) and post (week 32)
  Inflammatory biomarker
Vitamin D | pre (week 0) and post (week 32)
  Vitamin

SECONDARY OUTCOMES:
Glutamic-oxaloacetic transaminase (GOT) | pre (week 0) and post (week 32)
  Hepatic biomarker
Glutamic-pyruvic transaminase (GPT) | pre (week 0) and post (week 32)
  Hepatic biomarker
Gamma- glutamyl transpeptidase (GGT) | pre (week 0) and post (week 32)
  Hepatic biomarker
Alkaline phosphatase enzyme (ALP) | pre (week 0) and post (week 32)
  Hepatic biomarker
Systolic blood pressure (SBP) | pre (week 0) and post (week 32)
  Cardiovascular measure
Diastolic blood pressure (SBP) | pre (week 0) and post (week 32)
  Cardiovascular measure
Up and Go test (UGT) | pre (week 0) and post (week 32)
  Functional test
Age | pre (week 0) and post (week 32)
  Sample demographic description
Height | pre (week 0) and post (week 32)
  Sample demographic description
Weight | pre (week 0) and post (week 32)
  Sample demographic description
Body mass index (BMI) | pre (week 0) and post (week 32)
  Sample demographic description
Fat mass percentage (% fat mass) | pre (week 0) and post (week 32)
  Sample demographic description